CLINICAL TRIAL: NCT06207890
Title: An Analysis of Participation Trends: Observing Patient Engagement in Anorexia Nervosa Clinical Trials
Brief Title: Exploring Clinical Study Experiences of People With Anorexia Nervosa
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 58191532
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study seeks to delve into the firsthand experiences of patients diagnosed with anorexia nervosa who partake in a separate clinical trial featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

By joining this clinical trial, individuals have the unique opportunity to contribute to the betterment of future anorexia nervosa patients and play an active role in advancing medical research.

ELIGIBILITY:
Inclusion Criteria:

* Patient has self-identified as planning to enroll in a clinical trial
* Patient has been diagnosed with anorexia nervosa
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with anorexia nervosa who are actively considering enrolling in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in anorexia nervosa clinical trial | 3 months
Rate of patients who remain in anorexia nervosa clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walsh BT, Hagan KE, Lockwood C. A systematic review comparing atypical anorexia nervosa and anorexia nervosa. Int J Eat Disord. 2023 Apr;56(4):798-820. doi: 10.1002/eat.23856. Epub 2022 Dec 12. PMID 36508318
- [Background] Paolacci S, Kiani AK, Manara E, Beccari T, Ceccarini MR, Stuppia L, Chiurazzi P, Dalla Ragione L, Bertelli M. Genetic contributions to the etiology of anorexia nervosa: New perspectives in molecular diagnosis and treatment. Mol Genet Genomic Med. 2020 Jul;8(7):e1244. doi: 10.1002/mgg3.1244. Epub 2020 May 5. PMID 32368866
- [Background] Parpia R, Spettigue W, Norris ML. Approach to anorexia nervosa and atypical anorexia nervosa in adolescents. Can Fam Physician. 2023 Jun;69(6):387-391. doi: 10.46747/cfp.6906387. PMID 37315981

DOCUMENTS (1):
  • Informed Consent Form (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT06207890/ICF_000.pdf